CLINICAL TRIAL: NCT04099212
Title: OBSERVATIONAL CASE-ONLY PROSPECTIVE STUDY OF EFFECTIVENESS AND SAFETY OF 15% TOPICAL RESORCINOL FOR ADULTS WITH HURLEY I-II HIDRADENITIS SUPPURATIVA.
Brief Title: 15% TOPICAL RESORCINOL FOR HURLEY I-II HIDRADENITIS SUPPURATIVA.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-RES-2018-01
Record Dates: First submitted 2019-09-09; First posted 2019-09-23 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2019-04

CONDITIONS: HYDRADENITIS
Keywords: RESORCINOL; HIDRADENITIS SUPPURATIVA
MeSH Terms: conditions — Hidradenitis; Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Patients with HS I-II in monotherapy treatment of topical resorcinol 15%

SUMMARY:
Prospective, observational cross-sectional study to evaluate the response of patients with HS I-II to monotherapy treatment of topical resorcin 15%, taking into account its safety, impact on quality of life and subclinical evolution.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Diagnosed with HS Hurley I-II degree.
* Patients that have at least 1 or more swollen up nodules and/or abscess.
* Availability of affected region control ultrasound prior to resorcine treatment beginning.

Exclusion Criteria:

* Age < 18 years.
* Number of draining fistula above 20.
* Patients in active treatment with immunomodulators.
* Patients in active treatment with antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that suffer from Hs Hurley I-II from the Andalusian Public Health System that are been follow up by the Dermatology Unity of Clinical Management of the HUVM.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the change in the disease severity | Up to 16 weeks
  Score change in the Hidradenitis Sartorius modified score

SECONDARY OUTCOMES:
Usage profile | Initial
  Descriptive measurement of demographic and clinical variables (central tendency, dispersion and distribution of tendencies) prior to the start of treatment.
Evaluate the security of the treatment | Up to 16 weeks
  Number and description of adverse effects, analysing the percentage and frequency of withdrawal and treatment suspension due to side effects.
Evaluate the changes in the patient´s quailty of life due to the treatment | Up to 16 weeks
  Quantified by the average absolute change of the dermatology life quality index (DLQI) score, a questionnaire that measures the effect that the skin disease has on the quality of life of an affected person.
Evaluate the changes in the patient´s quailty of life due to the treatment 2 | Up to 16 weeks
  Quantified by the average absolute changein the visual analog scale of pain, odor and suppuration, a scale used to measure the intensity or frequency of the symptoms related to the pain, odor and suppuration of the disease.
Total and partial ultrasound responders frequency of distribution. | Up to 16 weeks
  Change in number of fistulas, pseudocysts and abscess as well as change in doppler activity.
  Defining total ultrasound responders as the ones that have a smaller number of pseudocysts, liquid collections, fistulas, smaller size and thickness of the main injury and less doppler activity than the registered in the baseline ultrasound and partial ultrasound responders as the ones that have less activity than in the baseline ultrasound in at least one of the previous variables without increase in any of the others.
Evaluate the frequency of responders | Up to 16 weeks
  Defining responder as the combination of the decrease in the abscess/nodule count by at least 50% (minimum of one), without increase in the number of draining fistulas and the number of abscesses.
Evaluate the change in the disease severity. | Up to 16 weeks
  Score change in the Physician Global Assesment scale for Supurative Hidradenitis

CONTACTS AND LOCATIONS:
Overall Officials: David Moreno Ramírez, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain